CLINICAL TRIAL: NCT07356206
Title: Between Paws and Affections: Impact of Dog Assisted Therapy on Pain, Emotional Symptoms, and Functioning in Fibromyalgia
Brief Title: Between Paws and Affections - Impact of Dog-Assisted Therapy in Fibromyalgia Patients
Acronym: IDAT26
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minho (Other)
Collaborators: Unidade Local de Saúde do Alto Ave, EPE (Other)
Responsible Party: Principal Investigator, Armando Almeida, Associate Professor, University of Minho
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REF.19/2024
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Fibromyalgia (FM)
Keywords: Fibromyalgia; Dog-Assisted Therapy; Pain; Anxiety; Depression; Psychoeducation and Relaxation; Fuctional Impact; Catastrophizing; follow-up evaluations; Hospital Anxiety and Depression Scale (HADS); Pain Catastrophizing Scale; Portuguese Fibromyalgia Impact Questionnaire (FIQ P); Numerical Rating Scale (NRS); adapted Wong Baker Faces Pain Scale; Portuguese Brief Pain Inventory - Short Form
MeSH Terms: conditions — Fibromyalgia; Pain; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral: Dog Assisted Therapy (DAT - "Between Paws and Affections") (Experimental): Intervention group that will receive a total of 10 group sessions at the Psychiatry Day Hospital of ULS Alto Ave, organized into 4 weekly structured sessions (combining psychoeducation on fibromyalgia and chronic pain, functional training and self care, lifestyle counseling and guided relaxation, all mediated by trained therapy dogs and a professional dog handler), followed by 6 monthly guided relaxation "booster" sessions with the dogs.
  Interventions: Behavioral: Behavioral: Dog Assisted Therapy (DAT - "Between Paws and Affections")
- Behavioral: Psychoeducation and Relaxation without Dogs (Control) (Active Comparator): New active control group that will receive the same 10-session program, with structure, duration, and content identical to the DAT arm (4 weekly structured psychoeducation and functional/self-care sessions plus 6 monthly guided relaxation "booster" sessions), but delivered entirely without dogs.
  Interventions: Behavioral: Behavioral: Psychoeducation and Relaxation without Dogs (Control)

INTERVENTIONS:
Behavioral: Behavioral: Dog Assisted Therapy (DAT - "Between Paws and Affections") — Dog Assisted Therapy (DAT - "Between Paws and Affections") - Intervention group that will receive a total of 10 group sessions at the Psychiatry Day Hospital of ULS Alto Ave, organized into 4 weekly structured sessions (combining psychoeducation on fibromyalgia and chronic pain, functional training and self care, lifestyle counseling and guided relaxation, all mediated by trained therapy dogs and a professional dog handler), followed by 6 monthly guided relaxation "booster" sessions with the dogs.
  Arms: Behavioral: Dog Assisted Therapy (DAT - "Between Paws and Affections")
Behavioral: Behavioral: Psychoeducation and Relaxation without Dogs (Control) — Control group that will receive the same 10 session program, with structure, duration and content identical to the DAT arm (4 weekly structured psychoeducation and functional/self care sessions plus 6 monthly guided relaxation "booster" sessions), but delivered entirely without dogs.
  Arms: Behavioral: Psychoeducation and Relaxation without Dogs (Control)

SUMMARY:
The purpose of this study is to evaluate the effectiveness and medium-term maintenance of a structured dog-assisted therapy (DAT) protocol, "Entre Patas e Afetos" (Between Paws and Affections), in reducing pain, anxiety and depressive symptoms and in improving functional status and quality of life in Portuguese patients with fibromyalgia (FM) followed at ULS Alto Ave, with systematic outcome assessment in the immediate post intervention phase (T2), 6-month follow-up (T3) and 12-month follow-up (T4).

DETAILED DESCRIPTION:
This is a prospective, non-randomized clinical trial with a control group, conducted at the Day Hospital of the Psychiatry and Mental Health Department of ULS Alto Ave, as an academic research project within a PhD in Medicine at the University of Minho.

The original pilot trial (Ref. 19/2024), including 34 women with FM, showed statistically significant improvements in maximum and average pain intensity, pain interference, total pain catastrophizing and its subscales (helplessness, magnification, rumination), anxiety (HADS) and functional impact (FIQ-P). However, depressive symptoms showed only a non-significant trend for improvement. Critically, analysis of 6-month follow-up data (T3) revealed partial erosion of the initial gains: pain intensity, pain interference, functional impact, and emotional symptoms showed variable maintenance patterns, with particular vulnerability to relapse in depressive symptoms, supporting the need for a prolonged intervention with maintenance sessions to consolidate gains and prevent deterioration over time.

The prolongation protocol comprises: (1) continuation of the initial control group with five monthly relaxation sessions; and (2) inclusion of a new intervention group receiving 10 DAT sessions (4 weekly structured dog-assisted therapy sessions plus 6 monthly guided-relaxation "booster" sessions with dogs) and a new active control group receiving an identical psychoeducational and relaxation program without dogs.

Sessions are group-based (up to 5 patients), last 60 minutes, and are delivered in a dedicated therapy room in the Psychiatry Day Hospital, by a multidisciplinary team (psychiatrist, psychologist, nurse, physiatrist) together with trained therapy dogs (Ari, Maica) and a professional dog handler, with appropriate veterinary follow-up and liability/health insurance.

Eligibility is assessed by a psychiatrist according to predefined inclusion and exclusion criteria; eligible patients provide written informed consent and complete baseline questionnaires (T1) up to four weeks before starting the intervention. Outcome assessments are performed immediately after session 4 (T2), at 6 months after session 4, and before session 10 (T3), and at 12 months after the end of the intervention (T4), in order to monitor the short-term response, the 6-month maintenance or progression of gains, and the 12-month trajectory associated with the monthly booster sessions. All procedures follow the previously approved protocol (Ref. 19/2024) and comply with the requirements of the institutional Ethics Committee and the Data Protection Officer, with no new data categories or processing purposes, and an addendum specifically for the extension of the study has been submitted and approved.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Confirmed diagnosis of fibromyalgia
* Being followed at ULS Alto Ave by the Multidisciplinary Pain Unit, Internal Medicine (Auto immune diseases), Physical and Rehabilitation Medicine or Neurology
* Ability to read and write Portuguese and to understand the study procedures
* Willingness and ability to participate voluntarily in the 10 session program and all scheduled assessments (T1-T4)
* Provision of written informed consent

Exclusion Criteria:

* Allergy to dogs or marked fear of dogs
* History of aggression towards animals
* History of oncological disease
* Concomitant systemic or rheumatologic disease that may confound pain and functional assessment
* Decompensated psychiatric disorder or severe cognitive impairment that may compromise comprehension of the protocol or adherence to the intervention
* Refusal to participate or withdrawal of consent at any point

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity (maximum and average) and pain interference | 13 months - From 1 month after enrollment to the end of treatment at 12 months after the first month
  Measured by the Portuguese Brief Pain Inventory - Short Form , at T2 (post session 4), T3 (6 month follow up) and T4 (12 month follow up), to capture both short term change and medium term maintenance at 6 and 12 months after the first month (T2). Self reported pain intensity using a Numeric Rating Scale with faces / adapted Wong Baker Faces Pain Scale, collected at each session to monitor pain fluctuations across the acute and maintenance phases.
Fibromyalgia impact and functional status | 13 months - From 1 month after enrollment to the end of treatment at 12 months after the first month
  Measured by the Portuguese Fibromyalgia Impact Questionnaire (FIQ P), at T2, T3 and T4, allowing evaluation of functional changes and their persistence at 6 and 12 months after the first month (T2)

SECONDARY OUTCOMES:
Anxiety and depressive symptoms | 13 months - From 1 month after enrollment to the end of treatment at 12 months after the first month
  Measured by the Hospital Anxiety and Depression Scale - Anxiety (HADS A, Portuguese version) and Depression (HADS D, Portuguese version) subscales, at T2, T3 and T4.
Pain catastrophizing | 13 months - From 1 month after enrollment to the end of treatment at 12 months after the first month
  (total score and subscales: helplessness, magnification, rumination), assessed by the Portuguese version of the Pain Catastrophizing Scale, at T2, T3 and T4, to explore whether reductions observed after 1 month of intervention (T2) are sustained or enhanced at 6 (T3) and 12 (T4) months.

CONTACTS AND LOCATIONS:
Overall Officials: Armando Almeida, Associate Professor, Study Chair — School of Medicine, University of Minho; Filipa Martins-Alves, Psychiatric Hospital Assistant, Principal Investigator — Psychiatry Department, Unidade Local de Saúde (ULS) Alto Ave
Locations (1):
- Unidade Local de Saúde (ULS) Alto Ave, Guimarães, Portugal

IPD SHARING:
Plan to Share IPD: No
Data protection in Portugal is very restricted concerning the sharing of patients' personal data.

REFERENCES:
- [Result] Meehan AG, Story DF, Medgett IC. Influence of the endothelium on the amplification by serotonin of vasoconstrictor responses to noradrenaline and sympathetic nerve stimulation in rabbit isolated ear artery. Eur J Pharmacol. 1987 Sep 23;141(3):339-46. doi: 10.1016/0014-2999(87)90550-4. PMID 3666031
- [Result] Yasuoka S, Nakayama T, Ishimi H, Ozaki T, Tsubura E, Ochi N. [Nephelometric immunoassay of albumin and IgG in bronchoalveolar lavage fluid (author's transl)]. Nihon Kyobu Shikkan Gakkai Zasshi. 1981 Apr;19(4):230-8. No abstract available. Japanese. PMID 7277909
- [Result] Nesbitt A, Heathcock R. Integration of hepatitis B vaccination into national immunisation programmes. Delivering vaccine to infants at risk is complex. BMJ. 1997 Jul 12;315(7100):121. doi: 10.1136/bmj.315.7100.121a. No abstract available. PMID 9240064
- [Result] Tokarski C. Coalition proposes Medicaid overhaul. Mod Healthc. 1989 Feb 24;19(8):3. No abstract available. PMID 10324920
- [Result] Danezis J. Antifertility agents and mammalian gonads. A proposal for assessing the effectiveness of antifertility compounds. Int J Fertil. 1968 Apr-Jun;13(2):95-102. No abstract available. PMID 5645535
- [Result] Ibekwe AO, Okoye BC. Subperiosteal mastoid abscesses in chronic suppurative otitis media. Ann Otol Rhinol Laryngol. 1988 Jul-Aug;97(4 Pt 1):373-5. doi: 10.1177/000348948809700408. PMID 3408111
- [Result] Rosado Mda L, Pereira JP, da Fonseca JP, Branco JC. [Cultural adaptation and validation of the "Fibromyalgia Impact Questionnaire"--Portuguese version]. Acta Reumatol Port. 2006 Apr-Jun;31(2):157-65. Portuguese. PMID 17058362
- [Result] Pais-Ribeiro J, Silva I, Ferreira T, Martins A, Meneses R, Baltar M. Validation study of a Portuguese version of the Hospital Anxiety and Depression Scale. Psychol Health Med. 2007 Mar;12(2):225-35; quiz 235-7. doi: 10.1080/13548500500524088. English, Portuguese. PMID 17365902
- [Result] Pandey RP, Himanshu; Gunjan; Mukherjee R, Chang CM. The Role of Animal-Assisted Therapy in Enhancing Patients' Well-Being: Systematic Study of the Qualitative and Quantitative Evidence. JMIRx Med. 2024 Mar 18;5:e51787. doi: 10.2196/51787. PMID 38606668
- [Result] Renner F, DeRubeis R, Arntz A, Peeters F, Lobbestael J, Huibers MJH. Exploring mechanisms of change in schema therapy for chronic depression. J Behav Ther Exp Psychiatry. 2018 Mar;58:97-105. doi: 10.1016/j.jbtep.2017.10.002. Epub 2017 Oct 6. PMID 29035800
- [Result] Malogiannis IA, Arntz A, Spyropoulou A, Tsartsara E, Aggeli A, Karveli S, Vlavianou M, Pehlivanidis A, Papadimitriou GN, Zervas I. Schema therapy for patients with chronic depression: a single case series study. J Behav Ther Exp Psychiatry. 2014 Sep;45(3):319-29. doi: 10.1016/j.jbtep.2014.02.003. Epub 2014 Feb 24. PMID 24650608
- [Result] Clark S, Martin F, McGowan RTS, Smidt J, Anderson R, Wang L, Turpin T, Langenfeld-McCoy N, Bauer B, Mohabbat AB. The Impact of a 20-Minute Animal-Assisted Activity Session on the Physiological and Emotional States in Patients With Fibromyalgia. Mayo Clin Proc. 2020 Nov;95(11):2442-2461. doi: 10.1016/j.mayocp.2020.04.037. Epub 2020 Aug 17. PMID 32819740
- [Result] Arnold LM, Bennett RM, Crofford LJ, Dean LE, Clauw DJ, Goldenberg DL, Fitzcharles MA, Paiva ES, Staud R, Sarzi-Puttini P, Buskila D, Macfarlane GJ. AAPT Diagnostic Criteria for Fibromyalgia. J Pain. 2019 Jun;20(6):611-628. doi: 10.1016/j.jpain.2018.10.008. Epub 2018 Nov 16. PMID 30453109
- See also: Azevedo LF, Costa-Pereira A, Mendonça L, Dias CC, Castro-Lopes JM. Tradução, adaptação cultural e validação do Inventário Resumido da Dor (Brief Pain Inventory - Short Form) para a população portuguesa. Dor. 2007;15(4):6-15 — https://www.aped-dor.org/socios/material_bibliografico/diversos_Questionarios_Dor-Rev_DOR_Volume15-n4-2007.pdf
- See also: Pereira MG, Machado JC, Alves S, et al. Adaptação e validação da versão portuguesa da Pain Catastrophizing Scale (PCS). Dor. 2017;25(1):16-25 — https://www.aped-dor.org/socios/material_bibliografico/diversos_EscalaCatastrofizacao_Dor-PCS.pdf
- See also: Oliveira AM, Batalha LMC, Fernandes AM, Gonçalves JC, Viegas RG. Uma análise funcional da Wong-Baker Faces Pain Rating Scale: linearidade, discriminabilidade e amplitude. Rev Enf Ref. 2014;IV(3):121-130 — http://dx.doi.org/10.12707/RIV14018
- See also: Direção-Geral da Saúde. Circular Normativa n.º 09/DGCG de 14/06/2003. Dor como 5º sinal vital - Registo sistemático da intensidade da Dor. Lisboa: DGS; 2003 — https://pns.dgs.pt/files/2015/08/Dor-como-5-Sinal-Vital-Registo-sistematico-da-intensidade-da-Dor.pdf